CLINICAL TRIAL: NCT04867369
Title: Pecs II Block Versus Surgeon Infiltration for Open Subpectoral Biceps Tenodesis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20-01978
Record Dates: First submitted 2021-04-28; First posted 2021-04-30 (Actual); Results first posted 2024-12-13 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Tendonitis
MeSH Terms: conditions — Tendinopathy | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Pecs II block (Experimental): 80 patients scheduled for open biceps tenodesis
  Interventions: Drug: Bupivacaine 20mL 0.5%; Drug: Bupivacaine 20mL 0.25%
- Surgical infiltration (Active Comparator): 80 patients scheduled for open biceps tenodesis
  Interventions: Drug: Bupivacaine 20mL 0.5%; Drug: Bupivacaine up to 15mL 0.25%

INTERVENTIONS:
Drug: Bupivacaine 20mL 0.5% — Interscalene nerve block with 20 mL 0.5% bupivacaine.
Drug: Bupivacaine 20mL 0.25% — Pecs II fascial plane block with 20 mL 0.25% bupivacaine.
  Arms: Pecs II block
Drug: Bupivacaine up to 15mL 0.25% — Local infiltration of 0.25% bupivacaine by the surgeon, up to 15 mL.
  Arms: Surgical infiltration

SUMMARY:
A phase IV, randomized, single-blind, single-center study measuring the effects of Pecs II block with 0.25% bupivacaine versus surgeon infiltration with 0.25% bupivacaine on postoperative pain control and opioid utilization in participants who undergo open subpectoral tenodesis.

ELIGIBILITY:
Inclusion Criteria:

1. Patients between 18 and 75 years of age
2. Patients undergoing shoulder arthroscopy with open subpectoral biceps tenodesis

Exclusion Criteria:

1. Patients younger than 18 and older than 75;
2. Patients with a history of chronic pain that have used opioids for pain management for 3 months or longer;
3. Patients who are allergic to oxycodone;
4. Patients with diagnosed or self-reported cognitive dysfunction;
5. Patients with a history of neurologic disorder that can interfere with pain sensation;
6. Patients with a history of drug or recorded alcohol abuse;
7. Patients who are unable to understand or follow instructions;
8. Patients with severe liver disease, renal insufficiency, congestive heart failure, and/or significant heart disease;
9. Patients with an allergy or contraindication to any of the medications used in the study, or patients with a contraindication to any study procedures;
10. Patients with a BMI over 45;
11. Any patient that the investigators feel cannot comply with all study related procedures;
12. NYU Langone Health students, residents, faculty or staff members.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2021-07-14 (Actual); Primary Completion 2023-11-08 (Actual); Study Completion 2023-11-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arthur Hertling, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset used in the published manuscript will be shared upon reasonable request beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research provided the investigator who proposes to use the data executes a data use agreement with NYU Langone Health. Requests may be directed to: Uchenna.Umeh@nyulangone.org. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required.
Access Criteria: Requests may be directed to Uchenna.Umeh@nyulangone.org.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pecs II Block | Surgical Infiltration
Started | 80 | 80
Completed | 79 | 80
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pecs II Block | Surgical Infiltration | Total
Number analyzed (Participants) | 79 | 80 | 159
Age, Continuous [Mean (Standard Deviation); unit: years] | 55 (11.78) | 55 (11.785) | 55 (11.783)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 35 | 63
  Male | 51 | 45 | 96
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 21 | 20 | 41
  Not Hispanic or Latino | 48 | 56 | 104
  Unknown or Not Reported | 10 | 4 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 2 | 3
  Asian | 5 | 3 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 11 | 16 | 27
  White | 32 | 37 | 69
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 30 | 22 | 52
Region of Enrollment [Number; unit: participants]
  United States | 79 | 80 | 159

OUTCOME MEASURES:

1. Primary Outcome: Opioid Utilization for the First 24 Hours After Surgery
Description: Opioid utilization is calculated as morphine milligram equivalents (MME); measurement includes opioid utilization during surgery.
Time Frame: Up to 24-Hours Post-Operation
Measure: Median (Inter-Quartile Range); unit: morphine milligram equivalents
Arm/Group | Pecs II Block | Surgical Infiltration
Number analyzed (Participants) | 80 | 80
morphine milligram equivalents | 17.5 [10.0 to 27.5] | 20 [10.0 to 30.0]

2. Secondary Outcome: Patient-reported Numerical Rating Scale (NRS) Score in Post Anesthesia Care Unit (PACU)
Description: In a Numerical Rating Scale (NRS), patients are asked to circle the number between 0 and 10; where 0 = no pain; and 10 = worst pain.
Time Frame: Typically 1-3 Hours Post-Operation
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Pecs II Block | Surgical Infiltration
Number analyzed (Participants) | 74 | 78
score on a scale | 0.5 [0.0 to 4.0] | 0 [0.0 to 2.0]

3. Secondary Outcome: Patient-reported Numerical Rating Scale (NRS) Score
Description: as for outcome 2
Time Frame: 24 Hours Post-Operation
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Pecs II Block | Surgical Infiltration
Number analyzed (Participants) | 66 | 60
score on a scale | 2.5 [0.0 to 6.0] | 3 [0.0 to 7.0]

4. Secondary Outcome: Patient-reported Numerical Rating Scale (NRS) Score
Description: as for outcome 2
Time Frame: Day 3 Post-Operation
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Pecs II Block | Surgical Infiltration
Number analyzed (Participants) | 60 | 55
score on a scale | 1.5 [0.0 to 5.0] | 3 [0.0 to 4.0]

5. Secondary Outcome: Number of Patients With Reactions to Surgical Subpectoral Incision - Movement
Description: Number of patients with movement during incision.
Time Frame: Intraoperative
Measure: Count of Participants; unit: Participants
Arm/Group | Pecs II Block | Surgical Infiltration
Number analyzed (Participants) | 75 | 80
Participants | 19 | 17

6. Secondary Outcome: Number of Patients With Reactions to Surgical Subpectoral Incision - Tachycardia
Description: Number of patients with tachycardia during incision.
Time Frame: Intraoperative
Measure: Count of Participants; unit: Participants
Arm/Group | Pecs II Block | Surgical Infiltration
Number analyzed (Participants) | 76 | 80
Participants | 14 | 19

7. Secondary Outcome: Number of Patients With Reactions to Surgical Subpectoral Incision - Sensation in Bicep
Description: Number of patients with sensation in bicep during incision.
Time Frame: Intraoperative
Measure: Count of Participants; unit: Participants
Arm/Group | Pecs II Block | Surgical Infiltration
Number analyzed (Participants) | 73 | 80
Participants | 30 | 32

ADVERSE EVENTS:
Time Frame: All events with start dates occurring any time after informed consent is obtained (baseline) until 7 (for non-serious AEs) or 30 days (for SAEs) after the last day of study participation, up to 34 days total.
Description: The study coordinator and PI were alerted if participants were admitted to the hospital. If they were admitted during the two week period, the PI determined if it was considered an adverse event related to the study.
Arm/Group | Pecs II Block | Surgical Infiltration
All-Cause Mortality (participants affected / at risk) | 0/80 | 0/80
Serious Adverse Events (participants affected / at risk) | 0/80 | 0/80
Other Adverse Events (participants affected / at risk) | 0/80 | 0/80

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-12-04): https://cdn.clinicaltrials.gov/large-docs/69/NCT04867369/Prot_SAP_000.pdf